CLINICAL TRIAL: NCT04374565
Title: Efficacy and Safety of High-Titer Anti-SARS-CoV-2 (COVID19) Convalescent Plasma for Hospitalized Patients With Infection Due to COVID-19 to Decrease Complications: A Phase II Trial
Brief Title: Convalescent Plasma for Treatment of COVID-19 Patients With Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jeffrey Sturek, MD, PhD, Assistant Professor of Pulmonary and Critical Care Medicine, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200114
Record Dates: First submitted 2020-04-27; First posted 2020-05-05 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Corona Virus Infection; SARS-CoV 2; SARS Pneumonia; Pneumonia
MeSH Terms: conditions — Coronavirus Infections; Pneumonia

STUDY DESIGN:
Intervention Model Description: This is a single arm phase II trial to assess preliminary efficacy and confirm safety of infusions of antiSARS-CoV-2 convalescent plasma in hospitalized patients with acute respiratory symptoms with or without confirmed interstitial COVID-19 pneumonia by CXR or chest CT. A total of 29 eligible subjects will be enrolled to receive high titer anti-SARS-CoV-2 plasma. Participants will be compared to a historical control group via retrospective chart review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study participants (Experimental): A total of 29 eligible subjects will be enrolled to receive high titer anti-SARS-CoV-2 plasma. Participants will be compared to a historical control group via retrospective chart review.
  Interventions: Drug: High-Titer Anti-SARS-CoV-2 (COVID 19) Convalescent Plasma

INTERVENTIONS:
Drug: High-Titer Anti-SARS-CoV-2 (COVID 19) Convalescent Plasma — Pathogen reduced SARS-CoV-2 convalescent plasma (1-2 units; ~200 mL each for a total of 200-400mls) given preferably in one day, but allowable to be given over 2 days if clinical circumstances delay infusions in 1 day), with titer to be determined after the unit has been infused.

SUMMARY:
This is a single arm phase II trial to assess efficacy and confirm safety of infusions of anti-SARS-CoV-2 convalescent plasma in hospitalized patients with acute respiratory symptoms,with or without confirmed interstitial COVID-19 pneumonia by chest Xray or CT. A total of 29 eligible subjects will be enrolled to receive anti-SARS-CoV-2 plasma.Outcomes will be compared to hospitalized controls with confirmed COVID-19 disease through retrospective chart review.

DETAILED DESCRIPTION:
There are no proven treatments for coronavirus disease (COVID-19) and associated pneumonia caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Recent experience in China suggests that convalescent immune plasma(CIP)may be an effective treatment for COVID-19. In the pandemic situation where there are no vaccines for COVID-19, specific antibodies in convalescent plasma induced by infection may provide passive protective immunity. Passive antibody therapy was the first immunotherapy dating back to the 1890's for the treatment of infectious diseases before the development of antibiotics 1940's. Experience from prior outbreaks with other coronaviruses, such as SARS-CoV-1 shows that such convalescent plasma contains neutralizing antibodies to the relevant virus. In SARS-CoV-2, passive antibody therapy from CIP probably provided protection by viral neutralization. CIP was also used in the 2013 Ebola epidemic. A small non-randomized study in Sierra Leone revealed a significant increase in survival for who received CIP4. CIP administration is the only approach that provides immediate immunity to patients who have been exposed or who have active disease.

This approach is immediately available from individuals who have recovered, are viral free,and can donate immune plasma (IP) containing high titer neutralizing antibodies. Passive antibody therapy can be given to a patient recently exposed or a patient who is developing an infection with COVID-19 by obtaining plasma units from immune individuals by standard plasmapheresis using FDA-approved blood banking procedures, cross matching the unit(s) to the recipients and infusing the unit(s) using standard transfusion procedures for blood products. Based on the safety and long-term experience with plasma infusions, plasma exchanges, and other procedures involving plasma or plasma product, this protocol was designed as a phase II single arm trial that involves the administration of antibodies to a given agent to a susceptible individual for the purpose of preventing or treating an infectious disease due to that agent.

The only antibody formulation that is available for emergent use is that found in convalescent plasma. As more individuals contract COVID-19 and recover, the number of potential donors will increase.

The principle of passive antibody therapy is that it is more effective when used for prophylaxis than for treatment of disease. When used for therapy, antibody is most effective when administered shortly after the onset of symptoms. The reason for temporal variation in efficacy is not well understood but could reflect that passive antibody works by neutralizing the initial inoculum, which is likely to be much smaller than that of established disease. Alternatively, antibodies may dampen the early inflammatory response leaving the infected individual asymptomatic. For example, antibody therapy for pneumococcal pneumonia was most effective when given shortly after the onset of symptoms and was of no benefit if antibody therapy was delayed beyond the third day of disease. For passive antibody therapy to be effective, a sufficient amount of antibody must be infused. The antibody will circulate in the blood, reach tissues,and provide protection against infection. Depending on the type of antibody, amount, and composition, the half-life can vary from weeks to months. It is under these circumstances, the investigators plan to treat patients who are sick enough to be hospitalized before the onset of overwhelming disease involving a systemic inflammatory response, sepsis, and/or ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Patients hospitalized with COVID-19 respiratory symptoms within 72 hours of admission to a"floor" bed (non-ICU bed) and confirmation via SARS-CoV-2 RT-PCR testing.
* Patient and/or surrogate is willing and able to provide written informed consent and comply with all protocol requirements.
* Patients with hematologic malignancies or solid tumors are eligible.
* Patients with autoimmune disorders are eligible.
* Patients with immunodeficiency and organ or stem cell transplant recipients are eligible.
* Patients who have received or are receiving hydroxychloroquine or chloroquine are eligible (but will be taken off the drug)
* Prior use of IVIG is allowed but the investigator should consider the potential for a hypercoagulable state.

Exclusion Criteria:

* Patients requiring mechanical ventilation or >6 liters per minute nasal cannula oxygen
* Patients on other anti-COVID-19 trials being treated with tocilizumab (anti-IL-6 receptor), Siltuximab (anti-IL-2), Remdesivir, or other pharmacological trials that may be initiated hereafter.
* A pre-existing condition or use of a medication that, in the opinion of the site investigator, may place the individual at a substantially increased risk of thrombosis (e.g., cryoglobulinemia, severe refractory hypertriglyceridemia, or clinically significant monoclonal gammopathy).
* Contraindication to transfusion or history of prior reactions to transfusion blood products.
* Medical conditions for which receipt of 500-600 mL of intravenous fluid may be dangerous to the subject (e.g., decompensated congestive heart failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Virginia Medical Center, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casadevall A, Scharff MD. Return to the past: the case for antibody-based therapies in infectious diseases. Clin Infect Dis. 1995 Jul;21(1):150-61. doi: 10.1093/clinids/21.1.150. PMID 7578724
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Zhang JS, Chen JT, Liu YX, Zhang ZS, Gao H, Liu Y, Wang X, Ning Y, Liu YF, Gao Q, Xu JG, Qin C, Dong XP, Yin WD. A serological survey on neutralizing antibody titer of SARS convalescent sera. J Med Virol. 2005 Oct;77(2):147-50. doi: 10.1002/jmv.20431. PMID 16121363
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Casadevall A, Pirofski LA. Antibody-mediated regulation of cellular immunity and the inflammatory response. Trends Immunol. 2003 Sep;24(9):474-8. doi: 10.1016/s1471-4906(03)00228-x. No abstract available. PMID 12967670
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Yeh KM, Chiueh TS, Siu LK, Lin JC, Chan PK, Peng MY, Wan HL, Chen JH, Hu BS, Perng CL, Lu JJ, Chang FY. Experience of using convalescent plasma for severe acute respiratory syndrome among healthcare workers in a Taiwan hospital. J Antimicrob Chemother. 2005 Nov;56(5):919-22. doi: 10.1093/jac/dki346. Epub 2005 Sep 23. PMID 16183666
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] China puts 245 COVID-19 patients on convalescent plasma therapy. In: Huaxia, (ed): XinhuaNet, 2020.
- [Background] Crowe JE Jr, Firestone CY, Murphy BR. Passively acquired antibodies suppress humoral but not cell-mediated immunity in mice immunized with live attenuated respiratory syncytial virus vaccines. J Immunol. 2001 Oct 1;167(7):3910-8. doi: 10.4049/jimmunol.167.7.3910. PMID 11564809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Participants
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Transferred to Intensive Care Unit (ICU)
Description: Will be done by comparing the admission rate to the ICU between patients who received convalescent plasma and a control group who did not enroll in the study, or receive another experimental therapy.
Time Frame: Days 0 - 60
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Participants | 4

2. Primary Outcome: 28 Day Mortality
Description: Will be done by comparing the 28 day mortality rate between enrolled subjects and the control group.
Time Frame: Days 0 - 28
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Participants | 2

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Will be collected from time of enrollment until completion of the study. The adverse events will be evaluated by CTCAE V5.0 and MedDRA.
Time Frame: Days 0 - 60
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Participants | 4

4. Secondary Outcome: Duration of SARS-CoV-2 Positivity
Description: Respiratory tract swabs will be collected on days, 0, 7, 14, and 21 and will be tested for SARS-CoV-2. The outcome measurement is determining the duration from date of infection until date of first documented negative PCR test, which was assed up to 21 days
Time Frame: Days 0 - 21
Measure: Mean (Standard Error); unit: days
Arm/Group | Study Participants
Number analyzed (Participants) | 29
days | 20.4 (1.57)

5. Secondary Outcome: Serum of Plasma Antibody Titer to SARS-CoV-2
Description: Serum or plasma will be collected and analyzed for SARS-CoV-2 antibody.
Time Frame: Day 28
Population: Median IgG anti-spoke protein (ug/ml)
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Study Participants
Number analyzed (Participants) | 29
ug/mL | 7.7 [0.1 to 112.1]

6. Secondary Outcome: Cellular and Humoral Immune Response
Description: Blood will be collected and analyzed for for Spike IgG levels.
Time Frame: Day 28
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Study Participants
Number analyzed (Participants) | 29
ug/mL | 58.0 [34.0 to 90.0]

7. Secondary Outcome: Supplemental Oxygen Free Days
Description: All days where a supplemental oxygen is needed will be recorded as a concomitant medication and will be subtracted from total days the participant is alive and enrolled in the study up to day 28 to determine the supplemental oxygen free days.
Time Frame: Days 0-28
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Days | 23.5 [21 to 26]

8. Secondary Outcome: Ventilator Free Days
Description: All days where a ventilator is needed will be recorded as a concomitant procedure and will be subtracted from total days the participant is alive and enrolled in the study up to day 28 to determine the ventilator free days.
Time Frame: Days 0 - 28
Measure: Mean (Standard Error); unit: days
Arm/Group | Study Participants
Number analyzed (Participants) | 29
days | 24.93 (1.46)

9. Secondary Outcome: ICU Free Days
Description: All days where the participant is admitted to the ICU will be recorded and subtracted from total days the participant is alive and enrolled in the study up to day 28 to determine the ICU free days.
Time Frame: Days 0 - 28
Measure: Mean (Standard Error); unit: days
Arm/Group | Study Participants
Number analyzed (Participants) | 29
days | 24.59 (1.61)

10. Secondary Outcome: Sequential Organ Failure Assessment Score Improvement
Description: Throughout the study, participants were evaluated by study physician using the sequential organ failure assessment score. This outcome measurement is looking for the number of participants who's score improved over the duration of the study.
Time Frame: days 0-28
Population: Number of participants whose score improved throughout their admission.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Participants | 27

11. Secondary Outcome: Number of Participants Who Needed for Vasopressors
Description: Concomitant medications will be recorded throughout the patients participation in the study and vasopressors will be recorded, if they are needed.
Time Frame: Days 0 - 60
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Participants | 4

12. Secondary Outcome: Number of Participants Who Needed Renal Replacement Therapy
Description: Renal function will be assessed throughout the patients participation in the study. If renal replacement therapy is needed, it will be captured as a concomitant procedure.
Time Frame: Days 0 - 60
Population: number of study patients who required renal therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Participants | 1

13. Secondary Outcome: Number of Participants Who Needed Extracorporeal Membrane Oxygenation (ECMO)
Description: Respiratory function will be assessed throughout the patients participation in the study. If ECMO is needed, it will be captured as a concomitant procedure.
Time Frame: Days 0 - 60
Population: number of patients who received ECMO
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Participants | 1

14. Secondary Outcome: Hospital Length of Stay (LOS)
Description: Will be calculated from the date the patient entered the hospital until they were discharged.
Time Frame: Days 0-60
Measure: Mean (Standard Error); unit: days
Arm/Group | Study Participants
Number analyzed (Participants) | 29
days | 9.39 (1.56)

15. Secondary Outcome: ICU LOS
Description: Will be calculated from the date the patient entered the ICU until they were discharged from the ICU.
Time Frame: days 0 - 60
Measure: Mean (Standard Error); unit: days
Arm/Group | Study Participants
Number analyzed (Participants) | 29
days | 2.93 (1.72)

16. Secondary Outcome: Number of Participants Who Had a Grade 3 or 4 Adverse Events (AEs)
Description: All adverse events will be recorded and evaluated by CTCAE v.5.0. All grade 3 and 4 AEs will be calculated to determine safety of convalescent plasma.
Time Frame: Adverse events were collected from day 0 to 7 days post infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 29
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day 0 to 7 days post infusion.
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 2/29
Serious Adverse Events (participants affected / at risk) | 4/29
Other Adverse Events (participants affected / at risk) | 11/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=29)
Sepsis (Blood and lymphatic system disorders) | 1 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=29)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension urgency (Cardiac disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 5 (6)
hypotension (Cardiac disorders) | 1 (1)
syncope (Vascular disorders) | 1 (1)
fever (Infections and infestations) | 3 (3)
epistaxis (General disorders) | 1 (1)
creatine increased (Hepatobiliary disorders) | 1 (1)
ALT/AST increased (Hepatobiliary disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT04374565/Prot_SAP_001.pdf